CLINICAL TRIAL: NCT02410993
Title: Current Treatment Strategy of Patients With Multivessel Disease or Left Main Coronary Artery Disease Indicated for Coronary Artery Bypass Graft Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0063
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CABG surgery: Candidates for CABG surgery for left main disease, three-vessel disease or two-vessel disease with proximal LAD stenosis indicated by current practice guideline
  Interventions: Procedure: CABG surgery

INTERVENTIONS:
Procedure: CABG surgery

SUMMARY:
According to 2011 ACCF/AHA guideline and 2014 ESC/EACTS guideline, CABG surgery was recommended for three-vessel coronary artery disease and left main coronary artery disease in the patients with stable ischemic heart disease as class I. 2-VD with proximal left anterior descending artery stenosis was also indicated for CABG surgery as class I recommendation. However, many patients have been recommended for PCI by catheterization laboratory cardiologist; 46% and 93% in the only-CABG candidates and both CABG and PCI candidates, retrospectively, defined by previous ACC/AHA guideline. Although the discordance between real practice in catheterization laboratory and guideline would be adjusted by recently updated guideline. The revascularization strategy for patients with 3-VD/LMD in real practice have been getting toward more PCI and less CABG surgery. In this study, we will identify the rate of CABG candidates who were treated with PCI or medical treatment instead of CABG surgery in different from current guideline. We are also going to compare two treatment strategies CABG surgery vs. PCI with 2nd generation DES regarding clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Left main disease, three-vessel disease or two-vessel disease with proximal LAD stenosis.

Exclusion Criteria:

* Previous PCI within 1 year
* Previous sternotomy
* Primary PCI for STEMI
* Contraindication or hypersensitivity to anti-platelet medications or contrast media
* Planned need for concomitant other cardiac surgery (eg, valve surgery or resection of aortic or left ventricular aneurysm, etc)
* Pregnant women or women with potential childbearing
* Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
* Inability to understand or read the informed content

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital-based, full-service hospitals with capability of both PCI and CABG surgery in addition to cardiac catheterization
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients treated with PCI or medical treatment despite of recommendation for CABG surgery | 1 month (After the revascularization strategy was finally decided)

SECONDARY OUTCOMES:
Reason of ineligibility for CABG surgery | 1 month (After the revascularization strategy was finally decided)
the composite of major cardiac and cerebrovascular event (MACCE) | 1 year follow up after revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea